CLINICAL TRIAL: NCT07296575
Title: A Multicenter Study on Multimodal Diagnosis and Process Optimization of Thyroid Diseases Based on Ultrasonic Intelligent Agents
Brief Title: Ultrasound Large-scale Model in Thyroid Field: A Multi-center Study on Medical-Engineering Integration
Status: Active, not recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: Zhejiang University (Other); First Affiliated Hospital of Gannan Medical University (Other); Ganzhou People's Hospital (Unknown); Tumor Hospital of Jiangxi Province (Unknown); Chudong Medical Group Hospital (Yugan County) (Unknown); Zhengzhou Third People's Hospital (Unknown); Xuzhou Hospital of Traditional Chinese Medicine (Unknown); Yifu Hospital Affiliated to Nanjing Medical University (Unknown); Fuyang people's hospital (Other); General Hospital of Ningxia Medical University (Other); Ji'an Central People's Hospital (Unknown); Harbin First Specialized Hospital (Unknown); Sun Yat-sen University (Other); Shanghai Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine (Unknown); Yancheng First People's Hospital (Other); Yangling Demonstration Zone Hospital of Shaanxi Province (Unknown); Beijing Friendship Hospital (Other); Fengfeng Mineral Bureau General Hospital of Hebei Province (Unknown); Hunan Provincial Tumor Hospital (Unknown); Pingdingshan first people's Hospital (Unknown); PLA Joint Logistics Support Force No. 908 Hospital (Unknown); Bai Cheng Central Hospital (Unknown); PLA Joint Logistics Support Force No. 901 Hospital (Unknown); the Affiliated Hospital of Jinggangshan University (Unknown); Ji'an Third People's Hospital (Unknown)
Responsible Party: Principal Investigator, Chunquan Zhang, Professor, Second Affiliated Hospital of Nanchang University
Other Study IDs: SecondNanchangU2025; IIT-O-2025-343 (Registry Identifier: Multicenter Study on Ultrasound-Guided Intelligent Thyroid Parathyroid Fusion Technology Integrating Medical and Engine)
Record Dates: First submitted 2025-12-07; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Thyroid Abnormalities; Thyroid; Thyroid Cancer
Keywords: thyroid; Artificial Intelligence; Ultrasound
MeSH Terms: conditions — Thyroid Diseases; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: No intervention — no Intervention

SUMMARY:
The goal of this observational study is to evaluate the diagnostic accuracy and clinical workflow integration of an ultrasound intelligent agent (UIA) for thyroid disease management in a real-world multicenter setting. The primary research question is:

Can the UIA improve diagnostic consistency and efficiency for thyroid nodules (TI-RADS 1-5), Hashimoto's thyroiditis, and cervical lymph node metastasis compared to traditional ultrasound interpretation? Participants will include adults (18-80 years) undergoing thyroid ultrasound at 16 participating hospitals across China. Key inclusion criteria cover patients with suspected thyroid disorders requiring imaging, while exclusion criteria address poor image quality or concurrent clinical trials. Over 2,000 cases (50% thyroid nodules, 30% diffuse lesions, 12.5% non-nodular abnormalities, 7.5% special populations) will be prospectively enrolled. Data collection integrates static/dynamic ultrasound images, laboratory results, and AI-generated reports. Primary endpoints include model performance metrics (AUC, sensitivity/specificity, TI-RADS Kappa ≥0.8), workflow efficiency (report generation time ≤5 minutes), and pediatric/pregnancy-specific reference standards. Secondary analyses will assess inter-rater reliability (Cohen's Kappa) and longitudinal outcomes via 6-12-month follow-up. This study aims to establish evidence-based guidelines for AI-augmented thyroid diagnosis, particularly in underserved regions, while addressing gaps in current AI validation frameworks related to multi-modality data fusion and special population adaptability.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-80, clinically suspected thyroid disease (e.g., enlargement, nodules, pain) requiring ultrasound examination;
* Diffuse lesions must demonstrate both ultrasound characteristics and laboratory evidence;
* Dynamic video must fully cover the maximum diameter of the nodule without significant probe movement;
* Voluntary signed informed consent.

Exclusion Criteria:

* Poor image quality (severe gas interference, artifacts obscuring structural visualization);
* Inability to cooperate with examination (consciousness impairment, extreme non-compliance);
* Prior participation in other thyroid ultrasound-related clinical trials; postoperative thyroid recurrence;
* Thyroid malformation/ectopia affecting visualization.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with clinically suspected thyroid abnormalities who have been prescribed a thyroid ultrasound examination
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive Performance of Large Models in Ultrasound Thyroid Applications for Thyroid Diseases | Within 12 months of enrollment for each patient at the time of study completion.
  Diagnosing thyroid diseases using a large model in the field of ultrasound thyroid imaging, with histopathological examination results of thyroid lesions as the gold standard, to evaluate the model's sensitivity, specificity, accuracy, and area under the receiver operating characteristic curve (AUC) for diagnosing thyroid diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tessler FN, Middleton WD, Grant EG, Hoang JK, Berland LL, Teefey SA, Cronan JJ, Beland MD, Desser TS, Frates MC, Hammers LW, Hamper UM, Langer JE, Reading CC, Scoutt LM, Stavros AT. ACR Thyroid Imaging, Reporting and Data System (TI-RADS): White Paper of the ACR TI-RADS Committee. J Am Coll Radiol. 2017 May;14(5):587-595. doi: 10.1016/j.jacr.2017.01.046. Epub 2017 Apr 2. PMID 28372962
- [Result] de Carlos J, Garcia J, Basterra FJ, Pineda JJ, Dolores Ollero M, Toni M, Munarriz P, Anda E. Interobserver variability in thyroid ultrasound. Endocrine. 2024 Aug;85(2):730-736. doi: 10.1007/s12020-024-03731-5. Epub 2024 Feb 19. PMID 38372907
- [Result] Patel J, Klopper J, Cottrill EE. Molecular diagnostics in the evaluation of thyroid nodules: Current use and prospective opportunities. Front Endocrinol (Lausanne). 2023 Feb 24;14:1101410. doi: 10.3389/fendo.2023.1101410. eCollection 2023. PMID 36909304
- See also: Guidelines for the Diagnosis and Treatment of Thyroid Nodules and Differentiated Thyroid Cancer — https://rs.yiigle.com/CN311282202303/1451011.htm
- See also: Thyroid Cancer Diagnosis and Treatment Guidelines — https://zhptwkxwx.cma-cmc.com.cn/CN/10.3877/cma.j.issn.1674-0793.2019.01.001